CLINICAL TRIAL: NCT06906640
Title: Implementation pRogram to Improve Screening and Management for CKD in Diabetes (Program 2) (IRIS-CKD)
Brief Title: Implementation pRogram to Improve Screening and Management for CKD in Diabetes (IRIS-CKD) (Program 2)
Acronym: IRIS-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry); Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00116493_1
Record Dates: First submitted 2025-02-21; First posted 2025-04-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease(CKD); Type 2 DM; Type 2 Diabetes Mellitus (T2DM)
Keywords: CKD; T2DM; T2D; Type 2 Diabetes; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: (IRIS-CKD Management Program) is a comparative effectiveness 1:1 randomized trial of two interventions (Management vs. Education) to improve implementation of GDMT for CKD in 420 patients with T2D. All potential participants will receive educational materials on importance and opportunities to treat CKD before randomization. After randomization, both Education and Management participants will receive targeted educational materials on CKD and GDMT. The primary outcome will be an opportunity score of CKD GDMT at 6 months based on prescriptions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (IRIS-CKD Management Program): Education (Active Comparator): Education: Participants will receive targeted educational materials related to their stage of CKD, including recommendations for potential GDMT to discuss with their primary care provider.
  Interventions: Other: (IRIS-CKD Management Program): Education
- (IRIS-CKD Management Program): GDMT (Active Comparator): Management: Participants will receive targeted educational materials, along with GDMT prescription, dose titration, and laboratory monitoring by a pharmacist/APP, as necessary, with guidance from a centralized algorithm and oversight from a nephrologist site PI.
  Interventions: Other: (IRIS-CKD Management Program): Education; Other: (IRIS-CKD Management Program): GDMT

INTERVENTIONS:
Other: (IRIS-CKD Management Program): Education — Patients randomized to the education arm will receive targeted education materials regarding their severity of CKD, including the potential for additional GDMT to slow CKD progression to discuss with their Primary Care Provider (PCP). At 6 months, the study pharmacist (or APP) will order repeat eGFR and UACR after 6 months to standardize CKD follow up during the study period.
Other: (IRIS-CKD Management Program): GDMT — Patients randomized to the education arm will receive targeted education materials regarding their severity of CKD, including the potential for additional GDMT to slow CKD progression to discuss with their PCP. At 6 months, the study pharmacist (or APP) will order repeat eGFR and UACR after 6 months to standardize CKD follow up during the study period. Plus, receive guided care by APP.
  Arms: (IRIS-CKD Management Program): GDMT

SUMMARY:
IRIS-CKD is a two-program implementation study to improve guideline-recommended screening and treatment of chronic kidney disease (CKD) in individuals with type 2 diabetes (T2D) in the United States.

DETAILED DESCRIPTION:
IRIS-CKD Management Program: will compare prescriptions for guideline-directed medical therapies (GDMT) during the study period. To account for variable GDMT requirements, we will use opportunity scores to compare intervention arms. Patients will be screened, identified and undergo consent by the study site. Patients will receive educational materials related to CKD screening in T2D and details regarding the testing intervention study as per site specific recruitment requirements. The primary objective is to determine whether implementing a guided management program versus education alone will improve prescription of GDMT for people with CKD and T2D. Patients will complete approximately 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (CKD Management)

  * Adults with type 2 diabetes (T2D)
  * Receiving primary care within the healthcare system, visit within 24 months (any PCP provider, including APP)
  * Evidence of CKD based on laboratory testing within the past 2 years (must be confirmed during screening if not checked within 3 months of enrollment):

    * UACR >300 mg/g or
    * eGFR <45 ml/min/1.73 m2 or
    * UACR ≥30 mg/g with eGFR <60 ml/min/1.73 m2
  * Receiving <100% GDMT at baseline. For patients with UACR <30 mg/g, GDMT includes sodium-glucose cotransporter-2 inhibitors (SGLT2i) therapy. For all other eligible patients, GDMT includes ACEi/ARB, SGLT2i, and Finerenone, unless contraindications for any of these therapies exist (e.g., hyperkalemia, diabetic ketoacidosis, etc.).

Exclusion Criteria:

* (CKD Management)

  * Type 1 diabetes
  * Most recent eGFR <20 ml/min/1.73 m2
  * Prior kidney transplant
  * Autosomal dominant polycystic kidney disease (ADPKD)
  * Active pregnancy or plans for conception within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
CKD GDMT Opportunity Score at 6 months | 6 months
  Opportunity score of GDMT prescriptions at 6 months that were missing at baseline.
  The score will include prescriptions for GDMT that are active at month 6 or the loss of an indication for the GDMT.

SECONDARY OUTCOMES:
CKD GDMT Opportunity Score at 6 months weighted by dose | 6 months
  Change in opportunity score from baseline to 6 months weighted by prescribed dose of GDMT.
CKD GDMT Opportunity Score at 3 months | 3 months
  Opportunity score of GDMT prescriptions at 3 months that were missing at baseline.
  The score will include prescriptions for GDMT that are active at month 3 or the loss of an indication for the GDMT.

OTHER OUTCOMES:
UACR change | 6 months
  Change in UACR after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neha Pagidipati, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No